CLINICAL TRIAL: NCT03710733
Title: Randomized Prospective Study of Accelerated Hypofractionated Whole Breast Irradiation Plus Sequential Boost Versus Concomitant Boost Following Breast Conservative Surgery
Brief Title: Accelerated Hypofractionated Whole Breast Irradiation Plus Sequential Boost Versus Concomitant Boost Following BCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Rimoun Ramsis Anis Boutrus, Lecturer of Radiation Oncology, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201617079.3
Record Dates: First submitted 2018-07-07; First posted 2018-10-18 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Radiotherapy Side Effect
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential boost (Active Comparator): Hypofractionated whole breast irradiation 40 Gy/15 fx (2.67 Gy/fx) plus sequential boost 10 Gy/4 fx (2.5 Gy/fx) to lumpectomy cavity
  Interventions: Radiation: Sequential boost
- Concomitant boost (Experimental): Hypofractionated whole breast irradiation 40 Gy/15 fx (2.67 Gy/fx) plus concomitant boost 8 Gy/15 fx (0.53 Gy/fx) to lumpectomy cavity
  Interventions: Radiation: Concomitant boost

INTERVENTIONS:
Radiation: Sequential boost — Boost (10 Gy/4 fx/1 week) is given after whole breast irradiation
  Arms: Sequential boost
Radiation: Concomitant boost — Boost (8 Gy/15 fx/3 weeks) is given with whole breast irradiation
  Arms: Concomitant boost

SUMMARY:
A prospective study comparing sequential versus concomitant radiotherapy boost in breast conservative therapy.

DETAILED DESCRIPTION:
This study is a prospective randomized non-inferiority trial of accelerated hypofractionated whole breast irradiation plus sequential boost versus concomitant boost after breast conservative surgery. It will be conducted on 124 patients who will be randomized using permuted blocks. The primary outcome measured is the cosmetic outcome, while secondary outcomes are patient satisfaction (using breast questionnaire), acute toxicity (using RTOG acute toxicity scoring criteria), and late toxicity (using RTOG late toxicity scoring criteria).

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven breast cancer resected by lumpectomy
* Female patient
* Invasive breast cancer
* Negative surgical margin
* Age < or equal 50 years, or high-grade irrespective of age
* Appropriate stage for protocol entry i.e. no metastasis
* Performance Status 0-2
* Hormone receptor status:

  1. ER/PR Known
  2. Borderline results are considered positive

Exclusion Criteria:

* Metastatic patients
* Paget's disease of nipple
* Non-epithelial breast malignancy e.g. sarcoma, lymphoma
* Unresected suspicious microcalcifications in the same or contralateral breast
* Pregnant women
* Inability to delineate lumpectomy cavity
* Psychiatric or addictive disorders rendering treatment or follow-up difficult

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Cosmetic Outcome | 1 year
  Rate the qualities of the treated breast as compared with the untreated breast using European Organization for Research and Treatment of Cancer (EORTC) Cosmetic Rating System

SECONDARY OUTCOMES:
Patient Satisfaction: Breast Questionnaire (Breast Q) | 1 year
  Using Breast Questionnaire (Breast Q)
Acute Toxicity (Breast Skin) | During treatment and up to 3 months after treatment
  Using Radiation Therapy Oncology Group (RTOG) Acute Radiation Morbidity Scoring Criteria
Late Toxicity (Breast Skin, Heart, Lungs) | 1 year
  Using Radiation Therapy Oncology Group (RTOG) Late Radiation Morbidity Scoring Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Medhat El Sebaie, MD, Study Director — National Cancer Institute, Egypt
Locations (1):
- National Cancer Institute, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] Whelan TJ, Levine M, Julian J, Kirkbride P, Skingley P. The effects of radiation therapy on quality of life of women with breast carcinoma: results of a randomized trial. Ontario Clinical Oncology Group. Cancer. 2000 May 15;88(10):2260-6. PMID 10820347
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] van der Laan HP, Dolsma WV, Maduro JH, Korevaar EW, Hollander M, Langendijk JA. Three-dimensional conformal simultaneously integrated boost technique for breast-conserving radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):1018-23. doi: 10.1016/j.ijrobp.2007.01.037. Epub 2007 Mar 26. PMID 17379440